CLINICAL TRIAL: NCT01676610
Title: Infant Pulse Oximetry in Pakistan (iPOP) Study: Utility and Feasibility of Integrating Pulse Oximetry Into the Routine Assessment of Young Infants at First-level Clinics in Karachi, Pakistan
Brief Title: Infant Pulse Oximetry in Pakistan Study
Acronym: iPOP
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Daniel Roth, Staff Physician, Paediatric Medicine, The Hospital for Sick Children
Other Study IDs: 1000028096
Record Dates: First submitted 2012-08-22; First posted 2012-08-31 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Hypoxemia; Neonatal Sepsis; Pneumonia
Keywords: Pulse Oximetry; Pediatrics; Pakistan; Hypoxemia; Neonatal Sepsis; Pneumonia
MeSH Terms: conditions — Hypoxia; Neonatal Sepsis; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infants presenting to the Clinic: Infants presenting to the Bilal and Bhains Colony Health Center. Devices used to measure Pulse Oximetry (PO) include Rad-5v by Masimo, TuffSat by GE, N-65 by Nellcor, PRO2 by Conmed, and Lifebox by Acare.

SUMMARY:
Hypoxemia is an abnormally low concentration of oxygen in the blood, and is an important sign of cardio-respiratory compromise in acutely ill patients. Pulse oximetry (PO) is a rapid, portable, non-invasive and accurate method of measuring arterial hemoglobin oxygenation (Sp02), and can therefore be readily implemented to detect hypoxemia in the clinical setting. In this research study, we propose to test the hypothesis that the use of pulse oximetry to detect hypoxemia by first-level health workers' in Karachi, Pakistan is useful and feasible for the identification of the infants most urgently in need of medical care. We will enroll 1,400 infants 0-59 days of age who present to one of two primary health centers in Karachi. Infants will undergo brief clinical assessment by a community health worker (CHW) based on the WHO/UNICEF Integrated Management of Neonatal and Child Illness (IMNCI) algorithm, assessment by two pulse oximetry devices, and examination by a physician. The primary outcomes include prevalence of hypoxemia, feasibility of PO (e.g., time to obtain measurement, number of infants for who repeat measurements are required), and concordance between paired measurements on separate devices.

ELIGIBILITY:
Inclusion Criteria:

* Infant presenting to the Bilal or Bhains PHC in Karachi, Pakistan
* Age 0 - 59 days

Exclusion Criteria:

* Clinic visit is for scheduled injectable antibiotic administration (e.g., SAT trial)

Ages: 1 Day to 59 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Young infants, aged 0-59 days.
Sampling Method: Non-Probability Sample
Enrollment: 3149 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Prevalence of hypoxemia | Over the duration of hopsital stay, on average 24 hours

SECONDARY OUTCOMES:
Validity of PO | Baseline, +2 hours
  Validity of PO for the detection of infant illness, in comparison to physician assessment.
Comparison of PO Measurements | Baseline, +2 hours
  Between-devices comparison of PO measurements
Operational Feasibility | Baseline, +2 hours
  Operational feasibility (time to obtain measurement, acceptance by caregivers, robustness of devices)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Roth, MD, Principal Investigator — The Hospital for Sick Children
Locations (2):
- The Hospital for Sick Children, Toronto, Ontario, Canada
- Aga Khan University, Karachi, Pakistan